CLINICAL TRIAL: NCT02730221
Title: Administrative Workload in the Intensive Care Unit (AWIC Study)
Brief Title: Administrative Workload in the Intensive Care Unit
Acronym: AWIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Angelique Spoelstra-de Man, Dr. A.M.E. Spoelstra--de Man, Amsterdam UMC, location VUmc
Other Study IDs: 2015.564
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Critical Illness
Keywords: Administrative workload; Patient data management system; Intensive Care Unit; Work sampling method; Nursing Activity Score
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients admitted during measurement 1: All patients admitted to the Intensive Care and Medium Care Unit during a two-week study period before the implementation of a new electronic patient data management system
- Patients admitted during measurement 2: All patients admitted to the Intensive Care and Medium Care Unit during a two-week study period after the implementation of a new electronic patient data management system

SUMMARY:
A prospective observational study in the Intensive Care Unit and the Medium Care Unit in a university hospital in Amsterdam. Recent studies show that administrative tasks occupy more than 30% of the workload. One-third of these administrative tasks is unrelated to care. The administrative workload of physicians and nurses will be observed and quantified using two different methods. The amount of time physicians and nurses are logged on into the patient data management system (PDMS) will be measured and the time spent on different work tasks will be monitored with a work sampling method. Two different patient data management systems will be compared.

DETAILED DESCRIPTION:
In recent years, regulatory authorities request a growing number of protocols and checklists to improve healthcare. Though the intention is to prevent medical mistakes and to improve patient care, these demands might result in an increased administrative workload for physicians and nurses. Recent studies show that administrative tasks and documentation occupy more than thirty percent of the workload of physicians, of which one-third is unrelated to care. This time spent on administration could lower the amount of time spent with the patient and the patient's family. In the Intensive Care Unit and the Medium Care Unit, most of the administrative tasks are executed within the patient data management system. The way an electronic patient data management system is set up could impact the administrative workload for physicians and nurses. A prospective observational study at the department of Intensive and Medium Care of the University medical centre will be performed with the aim to quantify the time spent on direct patient care versus administrative work. Two different patient data management systems will be compared at different points in time. The Nursing Activity Score and other patient characteristics will be registered for all the admitted patients during the two study periods.

The administrative workload of physicians and nurses will be measured before and after the implementation of a new patient data management system, using the following methods:

* Login time in the electronic patient data management system during fourteen consecutive days in the Intensive Care Unit and the Medium Care Unit
* Timing of activities of physicians and nurses with a work sampling method during five consecutive day shifts in the Intensive Care Unit

ELIGIBILITY:
Inclusion Criteria:

* Admission to the Intensive Care Unit during one of the two study periods

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to the Intensive Care Unit during one of the two study periods
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-05 (Actual); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Login time in the PDMS per hour for nurses | 24 hours a day
  The amount of time being logged on to the PDMS per hour will be calculated for different shifts
Login time in the PDMS per hour for doctors | 24 hours a day
  The amount of time being logged on to the PDMS per hour will be calculated for different shifts
Amount of time spent on administrative work and documentation per shift for nurses | 9 hours a day
  The amount of time spent on administrative tasks and documentation during dayshifts measured with a work sampling methode
Amount of time spent on administrative work and documentation per shift for doctors | 9 hours a day
  The amount of time spent on administrative tasks and documentation during dayshifts measured with a work sampling methode

SECONDARY OUTCOMES:
Amount of time spent on direct patient care per shift for nurses | 9 hours a day
  The amount of time spent on direct care during dayshifts measured with a work sampling methode
Amount of time spent on direct patient care per shift for doctors | 9 hours a day
  The amount of time spent on direct care during dayshifts measured with a work sampling methode

CONTACTS AND LOCATIONS:
Overall Officials: Angelique ME Spoelstra - de Man, MD PhD, Study Director — Amsterdam UMC, location VUmc
Locations (1):
- VUMedicalCentre, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li L, Hains I, Hordern T, Milliss D, Raper R, Westbrook J. What do ICU doctors do? A multisite time and motion study of the clinical work patterns of registrars. Crit Care Resusc. 2015 Sep;17(3):159-66. PMID 26282253
- [Background] Armstrong E, de Waard MC, de Grooth HJ, Heymans MW, Reis Miranda D, Girbes AR, Spijkstra JJ. Using Nursing Activities Score to Assess Nursing Workload on a Medium Care Unit. Anesth Analg. 2015 Nov;121(5):1274-80. doi: 10.1213/ANE.0000000000000968. PMID 26484461
- [Background] Bosman RJ. Impact of computerized information systems on workload in operating room and intensive care unit. Best Pract Res Clin Anaesthesiol. 2009 Mar;23(1):15-26. doi: 10.1016/j.bpa.2008.10.001. PMID 19449613
- [Background] Urden LD, Roode JI. Work sampling. A decision-making tool for determining resources and work redesign. J Nurs Adm. 1997 Sep;27(9):34-41. doi: 10.1097/00005110-199709000-00009. PMID 9300013
- [Background] Pelletier D, Duffield C. Work sampling: valuable methodology to define nursing practice patterns. Nurs Health Sci. 2003 Mar;5(1):31-8. doi: 10.1046/j.1442-2018.2003.00132.x. PMID 12603719
- [Background] Marasovic C, Kenney C, Elliott D, Sindhusake D. A comparison of nursing activities associated with manual and automated documentation in an Australian intensive care unit. Comput Nurs. 1997 Jul-Aug;15(4):205-11. PMID 9260381